CLINICAL TRIAL: NCT06443125
Title: Study on Therapeutic Mechanism of Natural Psychotherapy for Neurosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Yang Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Organization: Beijing HuiLongGuan Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASPsy6
Record Dates: First submitted 2023-09-26; First posted 2024-06-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; natural psychotherapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Natural Psychotherapy intervention for obsessive-compulsive disorder (Experimental): Inpatient naturopathic treatment was performed once a day for 45 consecutive days
  Interventions: Other: Natural psychotherapy

INTERVENTIONS:
Other: Natural psychotherapy — Draw ideas from traditional Chinese culture, learn from the practice of Morita therapy in Japan, and create local practice experience. At the same time, a variety of research methods such as cognitive assessment and brain imaging were used to establish the scientific, professional and objective evaluation indexes of the therapy.

SUMMARY:
explore objective indicators of the efficacy of natural psychotherapy in the treatment of disorders such as obsessive-compulsive disorder

DETAILED DESCRIPTION:
1. To evaluate the cognitive function, Cognitive control, emotion and other aspects of neurosis patients, and to understand and master the cognitive behavior indicators of this population.
2. Investigate the pathological mechanism of neurotic patients from the aspects of electroencephalic graph/functional magnetic resonance imaging (EEG/fMRI) and biology.
3. To investigate the therapeutic effect of natural psychotherapy on cognitive impairment and related mood, sleep and symptom intervention in neurotic patients. In order to achieve the symptoms of neurosis patients, cognitive impairment and related mood and sleep intervention and promotion, while providing a scientific basis for neurosis rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of obsessive-compulsive disorder or compulsive behavior
* Duration of symptoms for not less than 12 months
* Age 15-60 years old.
* You can participate in the whole experiment and offline assessment in Beijing

Exclusion Criteria:

* Documented disease of physical diseases including, but not limited to stroke, tumor, Parkinson's disease, Huntington's disease, seizure, epilepsy, history of brain trauma
* Subjects who suffered from alcohol or illegal drug abuse/dependence

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms | Baseline, 12 weeks
  Obsessive-compulsive symptoms were assessed according to the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), The total score ranges from 0 to 40, with higher scores indicating more severe symptoms.
Cognitive function | Baseline, 12 weeks
  Cognitive inhibition was assessed using the emotional color-word Stroop task. The emotional Stroop task is a type of being Widely used cognitive inhibition assessment tools. The longer the reaction time, the worse the cognitive inhibition ability.
Mood and behavior | Baseline, 12 weeks
  Mood changes judged using gait and face recognition
ERP components associated with cognitive function | Baseline, 12 weeks
  To explore the ERP component analysis related to cognitive inhibition and Behavioral inhibition in obsessive-compulsive disorder (OCD) by event related potential (ERP) analysis
rest fMRI in Obsessive-compulsive patients | Baseline, 12 weeks
  The changes of resting-state functional connectivity were analyzed in patients with OCD before and after intervention. Resting-state functional connectivity：FC(Functional connectivity). Resting-state functional brain imaging data were collected using a GE 3.0T magnetic resonance scanner (GE Discovery MR750) at the Brain Imaging Center, Institute of Psychology, Chinese Academy of Sciences.
Behavioral inhibition | Baseline, 12 weeks
  behavioral inhibition was assessed using the emotional stop signal task (SST). The emotional SST task is a type of being Widely used behavioral inhibition assessment tools. Among them, the greater the SSRT, the worse the behavioral inhibition ability.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang-Yang Zhang, M.D., Ph.D, Principal Investigator — Institute of Psychology, Chinese Academy of Science
Locations (2):
- China (2):
  - Anhui Mental Health Center, Hefei, Anhui
  - Institute of Psychology, Chinese Academy of Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No
Data with be available on request